CLINICAL TRIAL: NCT02107209
Title: Evaluation of Bronchoscopic Biological Lung Volume Reduction Therapy in Pulmonary Emphysema Patients
Brief Title: Low Cost Biological Lung Volume Reduction Therapy for Advanced Emphysema
Acronym: BLVR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mostafa Bakeer, Dr, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD68
Record Dates: First submitted 2014-04-02; First posted 2014-04-08 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Pulmonary Emphysema
MeSH Terms: conditions — Pulmonary Emphysema | interventions — Pneumonectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bronchoscopic Lung volume reduction using Autologous blood. (Experimental): Injection of 30 ml autologous blood plus 3ml calcium chloride plus 3 ml tranexamic acid per segment via fiber-optic bronchoscope
  Interventions: Procedure: Bronchoscopic Lung volume reduction
- Bronchoscopic Lung volume reduction using Fibrin glue (Active Comparator): injection of 30 ml locally prepared fibrin glue per segment via triple lumen balloon catheter passing through fiberoptic bronchoscopy
  Interventions: Procedure: Bronchoscopic Lung volume reduction

INTERVENTIONS:
Procedure: Bronchoscopic Lung volume reduction — Fiberoptic bronchoscopy is used to inject the biological agents into the targeted lung segment

SUMMARY:
The clinical utility of bronchoscopic methods for achieving lung volume reduction has been evaluated in patients with advanced emphysema because these procedures are uniformly safer than surgical volume reduction. These include one-way valves, or bronchial occlusive devices to collapse emphysematous regions of lung and bronchial fenestration with bypass stents to improve expiratory flow, wire coils implants that compress the airway and thermal vapor ablation that causes an acute injury with subsequent fibrosis and reductions in volume.

DETAILED DESCRIPTION:
Biologic lung volume reduction (BioLVR): it is a novel endobronchial approach, which uses a Biological agents aiming to reduce lung volume by blocking off the most emphysematous areas with a rapidly polymerizing sealant. The mechanism of action involves resorption atelectasis from airway occlusion, subsequent airspace inflammation, and then remodeling. This remodeling will lead to scarring that induces contraction of lung parenchyma and functional volume reduction can be expected within 6-8 weeks. Biological lung volume reduction occurs independent of the presence or absence of collateral ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Emphysema determined by HRCT of the chest with:

   * .Persistent symptoms (i.e. a baseline Modified Medical Research Council dyspnea (MRC) score of >2 despite medical therapy).
   * FEV1 /FVC < 70% and FEV1 20%-50 % (Sever and very sever airflow limitation according to GOLD 2013).
   * Hyperinflation (total lung capacity (TLC) > 110% pred and residual volume/total lung capacity (RV/TLC) > 120% pred.
2. Patients not candidate for or had refused lung volume reduction surgery.
3. Age > 40 yrs.

Exclusion Criteria:

1. Airflow limitation with FEV1 < 20%.
2. DLCO < 20%.
3. Current smoker.
4. Patients not candidate for FOB.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Post-procedure lung volume reduction | 12 week
  Change from the baseline high-resolution computed tomography (HRCT) volumetry Change from the baseline Residual Volume/Total Lung Capacity from baseline.

SECONDARY OUTCOMES:
Post-procedure Improvement in dyspnea and exercise capacity | 12 weeks
  Changes from the baseline post-bronchodilator forced expiratory volume at one second (FEV1) and forced vital capacity (FVC), diffusing capacity of lung for carbon monoxide (DLCO), six-minute walk distance (6MWD),modified medical research council (MMRC) dyspnea score.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Saad El-Morsi, Prof, Study Chair — Chest Medicine Department, Faculty of Medicine, Mansoura University
Locations (1):
- Chest Medicine Department, Faculty Of Medicine, Mansoura University, Al Mansurah, Al-dakahliya, Egypt